CLINICAL TRIAL: NCT01345019
Title: A Randomized, Double-Blind, Multicenter Study of Denosumab Compared With Zoledronic Acid in the Treatment of Bone Disease in Subjects With Newly Diagnosed Multiple Myeloma
Brief Title: Denosumab Compared to Zoledronic Acid in the Treatment of Bone Disease in Patients With Multiple Myeloma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Collaborators: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 20090482; 2010-020454-34 (EudraCT Number)
Record Dates: First submitted 2011-04-28; First posted 2011-04-29 (Estimated); Results first posted 2018-03-07 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Cancer; Hematologic Malignancies; Multiple Myeloma; Oncology; Bone Metastases; Multiple Myeloma Bone Lesions
Keywords: zoledronic acid; hematologic malignancies; SRE; skeletal-related event; blood cancer; lytic bone lesions; bone metastases; myeloma; fractures; spinal cord compression; radiation to bone; surgery to bone; bisphosphonates; Neoplasms, Plasma Cell; Paraproteinemias; Neoplasms; Neoplasm Metastasis; Bone Neoplasms; Bone Marrow Diseases; Blood Protein Disorders; Hematologic Diseases; multiple myeloma; denosumab; Neoplastic Processes; Bone Diseases; Diphosphonates; Bone Density Conservation Agents
MeSH Terms: conditions — Neoplasms; Hematologic Neoplasms; Multiple Myeloma; Neoplasms, Plasma Cell; Fractures, Bone; Spinal Cord Compression; Paraproteinemias; Neoplasm Metastasis; Bone Neoplasms; Bone Marrow Diseases; Blood Protein Disorders; Hematologic Diseases; Neoplastic Processes; Bone Diseases | interventions — Denosumab; Zoledronic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Zoledronic acid (Active Comparator): Zoledronic acid 4 mg intravenously plus placebo to denosumab subcutaniously (SC) once every 4 weeks (Q4W) in the double-blind treatment period (Since denosumab was determined to have a positive benefit:risk profile in the primary analysis of the study, per protocol, participants who were still undergoing Q4W scheduled assessments were offered open-label denosumab 120 mg SC Q4W for up to 2 years)
  Interventions: Drug: Zoledronic acid; Drug: Placebo to Denosumab; Drug: Denosumab (for the open-label treatment phase)
- Denosumab (Experimental): Denosumab 120 mg subcutaniously (SC) plus placebo to zoledronic acid intravenously once every 4 weeks (Q4W) in the double-blind treatment period (Since denosumab was determined to have a positive benefit:risk profile in the primary analysis of the study, per protocol, participants who were still undergoing Q4W scheduled assessments were offered open-label denosumab 120 mg SC Q4W for up to 2 years)
  Interventions: Drug: Denosumab; Drug: Placebo to zoledronic acid; Drug: Denosumab (for the open-label treatment phase)

INTERVENTIONS:
Drug: Denosumab — Administered by subcutaneous injection once every 4 weeks.
  Other Names: XGEVA®; AMG 162
  Arms: Denosumab
Drug: Zoledronic acid — Administered by intravenous infusion over 15 minutes once every 4 weeks
  Other Names: Zometa®
  Arms: Zoledronic acid
Drug: Placebo to Denosumab — Administered by subcutaneous injection once every 4 weeks.
  Arms: Zoledronic acid
Drug: Placebo to zoledronic acid — Administered by intravenous infusion over 15 minutes once every 4 weeks
  Arms: Denosumab
Drug: Denosumab (for the open-label treatment phase) — Administered by subcutaneous injection once every 4 weeks.
  Other Names: XGEVA®; AMG 162

SUMMARY:
The purpose of this study is to determine if denosumab is non-inferior to zoledronic acid in the treatment of bone disease from multiple myeloma.

ELIGIBILITY:
Inclusion Criteria:

* Documented evidence of multiple myeloma (per local assessment):
* Monoclonal plasma cells in the bone marrow greater than or equal to 10% and/or presence of a biopsy-proven plasmacytoma, and
* Monoclonal protein present in the serum and/or urine
* Radiographic (X-ray, or computer tomography [CT]) evidence of at least 1 lytic bone lesion (or at least 1 focal lesion per magnetic resonance imaging [MRI])
* Plan to receive or is receiving primary frontline anti-myeloma therapies
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2
* Age ≥ 18 years
* Adequate organ function, as defined by the following criteria (per central or local laboratory values):

  * Serum aspartate aminotransferase (AST) ≤ 2.0 x upper limit of normal (ULN)
  * Serum alanine aminotransferase ≤ (ALT) 2.0 x ULN
  * Serum total bilirubin ≤ 2.0 x ULN
  * Creatinine clearance ≥ 30 mL/min
  * Serum calcium or albumin-adjusted serum calcium 2.0 mmol/L (8.0 mg/dL) and 2.9 mmol/L (11.5 mg/dL)
* Written informed consent before any study-specific procedure is performed

Exclusion Criteria:

* Nonsecretory multiple myeloma based upon standard M-component criteria (ie, measurable serum/urine M-component) unless the baseline serum free light chain level is elevated
* POEMS syndrome (polyneuropathy, organomegaly, endocrinopathy, monoclonal protein, and skin changes)
* Plasma cell leukemia
* More than 30 days of previous treatment (before screening) with anti-myeloma therapy (does not include radiotherapy or a single short course of steroid [ie, less than or equal to the equivalent of dexamethasone 60 mg/day for 4 days]).
* Planned radiation therapy or surgery to the bone (does not include procedures performed before randomization)
* Prior administration of denosumab
* Use of oral bisphosphonates with a cumulative exposure of more than 1 year
* More than 1 previous dose of IV bisphosphonate administration
* Prior history or current evidence of osteonecrosis/osteomyelitis of the jaw
* Active dental or jaw condition which requires oral surgery, including tooth extraction
* Non-healed dental/oral surgery, including tooth extraction
* Planned invasive dental procedures
* Evidence of any of the following conditions per subject self-report or medical chart review:

  * Any prior invasive malignancy within 5 years before randomization
  * Any non-invasive malignancy not treated with curative intent or with knownactive disease within 5 years before randomization
  * Major surgery or significant traumatic injury occurring within 4 weeks before randomization
  * Active infection with Hepatitis B virus or Hepatitis C virus
  * Known infection with human immunodeficiency virus (HIV)
  * Active infection requiring IV anti-infective therapy
* Subject is pregnant or breast feeding, or planning to become pregnant within 5 months after end of treatment
* Female subject of child bearing potential is not willing to use highly effective contraception during treatment and for 5 months after the end of treatment (see section 6.3)
* Known sensitivity to any of the products to be administered during the study (eg, mammalian derived products, calcium or vitamin D)
* Subject is receiving or is less than 30 days since ending other experimental device or drug (no marketing authorization for any indication)
* Subject will not be available for follow-up assessment
* Any major medical or psychiatric disorder that in the opinion of the investigator, might prevent the subject from completing the study or interfere with the interpretation of the study results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1718 (Actual)
Dates: Start 2012-05-17 (Actual); Primary Completion 2016-07-19 (Actual); Study Completion 2019-03-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (262):
- United States (70):
  - Research Site, Tucson, Arizona
  - Research Site, Fayetteville, Arkansas
  - Research Site, Anaheim, California
  - Research Site, Campbell, California
  - Research Site, Encinitas, California
  - Research Site, Fresno, California
  - Research Site, Pleasant Hill, California
  - Research Site, Santa Barbara, California
  - Research Site, Santa Maria, California
  - Research Site, Stamford, Connecticut
  - Research Site, Washington D.C., District of Columbia
  - Research Site, Boynton Beach, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, Columbus, Georgia
  - Research Site, Savannah, Georgia
  - Research Site, Chicago, Illinois
  - Research Site, Joliet, Illinois
  - Research Site, Maywood, Illinois
  - Research Site, Niles, Illinois
  - Research Site, Skokie, Illinois
  - Research Site, Anderson, Indiana
  - Research Site, Fort Wayne, Indiana
  - Research Site, Indianapolis, Indiana
  - Research Site, Ames, Iowa
  - Research Site, Iowa City, Iowa
  - Research Site, Paducah, Kentucky
  - Research Site, New Orleans, Louisiana
  - Research Site, Scarborough, Maine
  - Research Site, Baltimore, Maryland
  - Research Site, Bethesda, Maryland
  - Research Site, Westminster, Maryland
  - Research Site, Boston, Massachusetts
  - Research Site, Danvers, Massachusetts
  - Research Site, Fairhaven, Massachusetts
  - Research Site, Detroit, Michigan
  - Research Site, Lansing, Michigan
  - Research Site, Jackson, Mississippi
  - Research Site, Springfield, Missouri
  - Research Site, Billings, Montana
  - Research Site, Lincoln, Nebraska
  - Research Site, Omaha, Nebraska
  - Research Site, North Las Vegas, Nevada
  - Research Site, Hackensack, New Jersey
  - Research Site, Lake Success, New York
  - Research Site, New York, New York
  - Research Site, Rochester, New York
  - Research Site, Fayetteville, North Carolina
  - Research Site, Goldsboro, North Carolina
  - Research Site, High Point, North Carolina
  - Research Site, Bismarck, North Dakota
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Hershey, Pennsylvania
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, West Reading, Pennsylvania
  - Research Site, Charleston, South Carolina
  - Research Site, Greenville, South Carolina
  - Research Site, Aberdeen, South Dakota
  - Research Site, Rapid City, South Dakota
  - Research Site, Sioux Falls, South Dakota
  - Research Site, Watertown, South Dakota
  - Research Site, Memphis, Tennessee
  - Research Site, Houston, Texas
  - Research Site, Lubbock, Texas
  - Research Site, Salt Lake City, Utah
  - Research Site, Christiansburg, Virginia
  - Research Site, Spokane, Washington
  - Research Site, Tacoma, Washington
  - Research Site, Morgantown, West Virginia
  - Research Site, Minocqua, Wisconsin
  - Research Site, Wauwatosa, Wisconsin
- Australia (10):
  - Research Site, Liverpool, New South Wales
  - Research Site, Tweed Heads, New South Wales
  - Research Site, Douglas, Queensland
  - Research Site, South Brisbane, Queensland
  - Research Site, Hobart, Tasmania
  - Research Site, Clayton, Victoria
  - Research Site, Epping, Victoria
  - Research Site, Malvern, Victoria
  - Research Site, Parkville, Victoria
  - Research Site, Prahran, Victoria
- Austria (6):
  - Research Site, Graz
  - Research Site, Innsbruck
  - Research Site, Krems
  - Research Site, Salzburg
  - Research Site, Vienna
  - Research Site, Wels
- Bulgaria (4):
  - Research Site, Pleven
  - Research Site, Plovdiv
  - Research Site, Sofia
  - Research Site, Varna
- Canada (13):
  - Research Site, Burnaby, British Columbia
  - Research Site, Winnipeg, Manitoba
  - Research Site, Moncton, New Brunswick
  - Research Site, St. John's, Newfoundland and Labrador
  - Research Site, Barrie, Ontario
  - Research Site, Newmarket, Ontario
  - Research Site, Sault Ste. Marie, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Windsor, Ontario
  - Research Site, Laval, Quebec
  - Research Site, Montreal, Quebec
  - Research Site, Québec, Quebec
  - Research Site, Trois-Rivières, Quebec
- Czechia (4):
  - Research Site, Brno
  - Research Site, Ostrava-Poruba
  - Research Site, Pilsen
  - Research Site, Prague
- France (19):
  - Research Site, Amiens
  - Research Site, Avignon
  - Research Site, Créteil
  - Research Site, Le Kremlin-Bicêtre
  - Research Site, Le Mans
  - Research Site, Lille
  - Research Site, Lyon Cédex 3
  - Research Site, Marseille
  - Research Site, Nantes
  - Research Site, Nice
  - Research Site, Paris
  - Research Site, Pessac
  - Research Site, Pierre-Bénite
  - Research Site, Pontoise
  - Research Site, Reims
  - Research Site, Rouen
  - Research Site, Saint-Quentin
  - Research Site, Strasbourg
  - Research Site, Villefranche-sur-Saône
- Germany (9):
  - Research Site, Bonn
  - Research Site, Chemnitz
  - Research Site, Cologne
  - Research Site, Essen
  - Research Site, Hamburg
  - Research Site, Kassel
  - Research Site, Leipzig
  - Research Site, Münster
  - Research Site, Regensburg
- Greece (5):
  - Research Site, Athens
  - Research Site, Heraklion
  - Research Site, Pátrai
  - Research Site, Piraeus
  - Research Site, Thessaloniki
- Hong Kong (2):
  - Research Site, Hong Kong
  - Research Site, New Territories
- Hungary (6):
  - Research Site, Budapest
  - Research Site, Debrecen
  - Research Site, Győr
  - Research Site, Gyula
  - Research Site, Kaposvár
  - Research Site, Szeged
- Ireland (3):
  - Research Site, Dublin
  - Research Site, Limerick
  - Research Site, Tullamore
- Italy (19):
  - Research Site, Ancona
  - Research Site, Bari
  - Research Site, Brescia
  - Research Site, Busto Arsizio
  - Research Site, Catania
  - Research Site, Florence
  - Research Site, Genova
  - Research Site, Messina
  - Research Site, Milan
  - Research Site, Napoli
  - Research Site, Novara
  - Research Site, Palermo
  - Research Site, Pescara
  - Research Site, Pisa
  - Research Site, Roma
  - Research Site, Rozzano MI
  - Research Site, Torino
  - Research Site, Udine
  - Research Site, Vimercate MB
- Japan (18):
  - Research Site, Nagoya, Aichi-ken
  - Research Site, Akita, Akita
  - Research Site, Kamogawa-shi, Chiba
  - Research Site, Fukuoka, Fukuoka
  - Research Site, Gifu, Gifu
  - Research Site, Ogaki-shi, Gifu
  - Research Site, Maebashi, Gunma
  - Research Site, Shibukawa-shi, Gunma
  - Research Site, Fukuyama-shi, Hiroshima
  - Research Site, Kobe, Hyōgo
  - Research Site, Kumamoto, Kumamoto
  - Research Site, Kyoto, Kyoto
  - Research Site, Okayama, Okayama-ken
  - Research Site, Kawagoe-shi, Saitama
  - Research Site, Tokushima, Tokushima
  - Research Site, Shibuya-ku, Tokyo
  - Research Site, Shinjuku-ku, Tokyo
  - Research Site, Toyama, Toyama
- Lithuania (2):
  - Research Site, Kaunas
  - Research Site, Vilnius
- Malaysia (4):
  - Research Site, Ipoh, Perak
  - Research Site, George Town, Pulau Pinang
  - Research Site, Kuching, Sarawak
  - Research Site, Ampang
- New Zealand (2):
  - Research Site, Christchurch
  - Research Site, Grafton, Auckland
- Poland (6):
  - Research Site, Legnica
  - Research Site, Lublin
  - Research Site, Słupsk
  - Research Site, Torun
  - Research Site, Warsaw
  - Research Site, Wroclaw
- Portugal (5):
  - Research Site, Braga
  - Research Site, Coimbra
  - Research Site, Lisbon
  - Research Site, Matosinhos Municipality
  - Research Site, Porto
- Russia (11):
  - Research Site, Dzerzhinsk
  - Research Site, Moscow
  - Research Site, Nizhny Novgorod
  - Research Site, Novosibirsk
  - Research Site, Penza
  - Research Site, Petrozavodsk
  - Research Site, Saint Petersburg
  - Research Site, Samara
  - Research Site, Saratov
  - Research Site, Volgograd
  - Research Site, Yekaterinburg
- Research Site, Singapore, Singapore
- Slovakia (3):
  - Research Site, Bratislava
  - Research Site, Nitra
  - Research Site, Nové Zámky
- South Korea (7):
  - Research Site, Anyang
  - Research Site, Busan
  - Research Site, Daegu
  - Research Site, Daejeon
  - Research Site, Gwangju
  - Research Site, Incheon
  - Research Site, Seoul
- Spain (9):
  - Research Site, Seville, Andalusia
  - Research Site, Palma de Mallorca, Balearic Islands
  - Research Site, Donostia / San Sebastian, Basque Country
  - Research Site, Salamanca, Castille and León
  - Research Site, Badalona, Catalonia
  - Research Site, Barcelona, Catalonia
  - Research Site, Ourense, Galicia
  - Research Site, Valencia, Valencia
  - Research Site, Madrid
- Switzerland (2):
  - Research Site, Chur
  - Research Site, Zurich
- Taiwan (6):
  - Research Site, Changhua
  - Research Site, Kaohsiung City
  - Research Site, Taichung
  - Research Site, Tainan
  - Research Site, Taipei
  - Research Site, Taoyuan District
- Turkey (Türkiye) (4):
  - Research Site, Adana
  - Research Site, Ankara
  - Research Site, Istanbul
  - Research Site, Izmir
- Ukraine (7):
  - Research Site, Cherkasy
  - Research Site, Dnipropetrovsk
  - Research Site, Ivano-Frankivsk
  - Research Site, Khmelnitskiy
  - Research Site, Kyiv
  - Research Site, Lviv
  - Research Site, Poltava
- United Kingdom (5):
  - Research Site, Harrow
  - Research Site, Inverness
  - Research Site, Leeds
  - Research Site, London
  - Research Site, Oxford

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication (or other new use) have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors, and if not approved, may be further arbitrated by a Data Sharing Independent Review Panel. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the link below.
URL: https://www.amgen.com/datasharing

REFERENCES:
- [Background] Raje N, Roodman GD, Willenbacher W, Shimizu K, Garcia-Sanz R, Terpos E, Kennedy L, Sabatelli L, Intorcia M, Hechmati G. A cost-effectiveness analysis of denosumab for the prevention of skeletal-related events in patients with multiple myeloma in the United States of America. J Med Econ. 2018 May;21(5):525-536. doi: 10.1080/13696998.2018.1445634. Epub 2018 Mar 5. PMID 29480139
- [Background] Raje N, Terpos E, Willenbacher W, Shimizu K, Garcia-Sanz R, Durie B, Legiec W, Krejci M, Laribi K, Zhu L, Cheng P, Warner D, Roodman GD. Denosumab versus zoledronic acid in bone disease treatment of newly diagnosed multiple myeloma: an international, double-blind, double-dummy, randomised, controlled, phase 3 study. Lancet Oncol. 2018 Mar;19(3):370-381. doi: 10.1016/S1470-2045(18)30072-X. Epub 2018 Feb 9. PMID 29429912
- [Background] Huang SY, Yoon SS, Shimizu K, Chng WJ, Chang CS, Wong RS, Gao S, Wang Y, Gordon SW, Glennane A, Min CK. Denosumab Versus Zoledronic Acid in Bone Disease Treatment of Newly Diagnosed Multiple Myeloma: An International, Double-Blind, Randomized Controlled Phase 3 Study-Asian Subgroup Analysis. Adv Ther. 2020 Jul;37(7):3404-3416. doi: 10.1007/s12325-020-01395-x. Epub 2020 Jun 10. PMID 32524500
- [Background] Terpos E, Raje N, Croucher P, Garcia-Sanz R, Leleu X, Pasteiner W, Wang Y, Glennane A, Canon J, Pawlyn C. Denosumab compared with zoledronic acid on PFS in multiple myeloma: exploratory results of an international phase 3 study. Blood Adv. 2021 Feb 9;5(3):725-736. doi: 10.1182/bloodadvances.2020002378. PMID 33560384
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 259 centers across 29 countries in Europe, North America, Asia, Australia/New Zealand, and Japan. Participants were enrolled from 17 May 2012 to 29 March 2016.
Pre-assignment Details: Randomization was stratified according to:
  * intent to undergo autologous peripheral blood stem cell (PBSC) transplantation
  * the antimyeloma agent being utilized/planned to be utilized in first-line therapy
  * stage (International Staging System [ISS]) at diagnosis
  * previous SRE (yes or no)
  * region (Japan yes or no)
Groups:
- Zoledronic Acid: Participants randomized to receive zoledronic acid 4 mg intravenously plus placebo to denosumab subcutaneously (SC) once every 4 weeks (Q4W) in the double-blind treatment phase. In the open-label treatment phase, remaining participants received denosumab 120 mg SC Q4W.
- Denosumab: Participants randomized to receive denosumab 120 mg subcutaneously (SC) plus placebo to zoledronic acid intravenously once every 4 weeks (Q4W) in the double-blind treatment phase. In the open-label treatment phase, remaining participants received denosumab 120 mg SC Q4W.
Period: Blinded Treatment Phase
Arm/Group | Zoledronic Acid | Denosumab
Started | 859 | 859
Received Treatment | 852 | 850
Completed (Still on-study as of blinded treatment analysis cutoff date of 05 January 2017) | 541 | 555
Not Completed | 318 | 304
Not completed — Death | 147 | 137
Not completed — Withdrawal by Subject | 103 | 112
Not completed — Completed Survival Follow-up | 21 | 9
Not completed — Disease Progression | 12 | 10
Not completed — Adverse Event | 6 | 13
Not completed — Administrative Decision | 10 | 8
Not completed — Noncompliance | 5 | 3
Not completed — Ineligibility Determined | 1 | 6
Not completed — Protocol Deviation | 5 | 0
Not completed — Other, Not Specified | 2 | 3
Not completed — Lost to Follow-up | 6 | 3
Period: Open Label Treatment Phase
Arm/Group | Zoledronic Acid | Denosumab
Started | 418 | 426
Completed | 227 | 233
Not Completed | 191 | 193
Not completed — Death | 49 | 48
Not completed — Withdrawal by Subject | 49 | 47
Not completed — Adverse Event | 30 | 51
Not completed — Administrative Decision | 30 | 15
Not completed — Disease Progression | 17 | 18
Not completed — Noncompliance | 5 | 4
Not completed — Lost to Follow-up | 1 | 2
Not completed — Pregnancy | 1 | 0
Not completed — Other, Not Specified | 9 | 7
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Zoledronic Acid: Participants randomized to receive zoledronic acid 4 mg intravenously plus placebo to denosumab subcutaneously once every 4 weeks in the double-blind treatment phase.
- Denosumab: Participants randomized to receive denosumab 120 mg subcutaneously plus placebo to zoledronic acid intravenously once every 4 weeks in the double-blind treatment phase.
- Total: Total of all reporting groups
Arm/Group | Zoledronic Acid | Denosumab | Total
Number analyzed (Participants) | 859 | 859 | 1718
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.3 (10.5) | 63.5 (10.6) | 63.4 (10.6)
Age, Customized [Count of Participants; unit: Participants]
  < 65 years | 464 | 472 | 936
  ≥ 65 years | 395 | 387 | 782
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 386 | 397 | 783
  Male | 473 | 462 | 935
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 35 | 35 | 70
  Not Hispanic or Latino | 819 | 823 | 1642
  Unknown or Not Reported | 5 | 1 | 6
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 699 | 711 | 1410
  Asian | 101 | 107 | 208
  Black or African American | 36 | 29 | 65
  Other | 19 | 10 | 29
  American Indian or Alaska Native | 3 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Multiracial | 0 | 1 | 1
  Missing | 1 | 0 | 1
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants] — A scale to assess a patient's disease status. 0 = Fully active, able to carry out all pre-disease performance without restriction; 1 = Restricted in physically strenuous activity, ambulatory and able to carry out work of a light nature; 2 = Ambulatory and capable of all self-care, unable to carry out any work activities. Up and about > 50% of waking hours; 3 = Capable of only limited self-care, confined to bed or chair > 50% of waking hours; 4 = Completely disabled, confined to bed or chair; 5 = Dead.
  Participants
    0 (Fully active) | 259 | 263 | 522
    1 (Restricted but ambulatory) | 413 | 400 | 813
    2 (Ambulatory but unable to work) | 187 | 196 | 383
Skeletal Related Event History [Number; unit: participants]
  Any Skeletal Related Event | 577 | 567 | 1144
  Pathological fracture | 463 | 479 | 942
  Spinal cord compression | 115 | 92 | 207
  Radiation therapy to bone | 139 | 118 | 257
  Surgery to bone | 144 | 142 | 286
Summary of Randomization Stratifications [Number; unit: participants] — Randomization was stratified by
  * Intent to undergo autologous peripheral blood stem cell (PBSC) transplantation: yes or no
  * The anti-myeloma agent being utilized/planned to be utilized in first-line therapy: novel therapy (included bortezomib, lenalidomide, or thalidomide) based or non-novel therapy-based,
  * International Staging System (ISS) stage at diagnosis: I (serum β2 microglobulin < 3.5 mg/L; serum albumin ≥ 3.5 g/dL) or II (neither stage I or III) or III (serum β2 microglobulin ≥ 5.5 mg/L),
  * Previous skeletal-related event (SRE): yes or no,
  * Region (Japan, non-Japan).
  participants
    Intent to undergo PBSC transplantation: Yes | 465 | 465 | 930
    Intent to undergo PBSC transplantation: No | 394 | 394 | 788
    Anti-myeloma agent utilized/planned: Novel | 821 | 819 | 1640
    Anti-myeloma agent utilized/planned: Non-novel | 38 | 40 | 78
    ISS stage at diagnosis: I | 268 | 263 | 531
    ISS stage at diagnosis: II | 313 | 319 | 632
    ISS stage at diagnosis: III | 278 | 277 | 555
    Previous SRE : Yes | 484 | 481 | 965
    Previous SRE : No | 375 | 378 | 753
    Region: Japan | 18 | 24 | 42
    Region: Non-Japan | 841 | 835 | 1676

OUTCOME MEASURES:

1. Primary Outcome: Time to First On-study Skeletal Related Event
Description: A skeletal-related event (SRE) is defined as one of the following: pathologic fracture (vertebral or non-vertebral), radiation therapy to bone (including the use of radioisotopes), surgery to bone, or spinal cord compression. Time to first on-study SRE is defined as the time interval (in days) from the randomization date to the date of first occurrence of on-study SRE. If there was no known event, and the participant was monitored for any one of the four SRE components, time to first on-study SRE was censored at the end of the treatment phase date or the primary analysis data cut-off date, whichever came first.
Time Frame: From randomization until the primary analysis data cut-off date of 19 July 2016 (per protocol); median time on study was 17.6 and 17.3 months in each treatment group respectively.
Population: All randomized participants
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Zoledronic Acid | Denosumab
Number analyzed (Participants) | 859 | 859
days | 730.0 [504.0 to 1014.0] | 695.0 [448.0 to NA] — Could not be estimated due to the low number of events
Statistical Analysis 1: Comparison: Zoledronic Acid vs Denosumab; Test type: Non-Inferiority — A two-stage approach was used for the non-inferiority test. First, the fixed margin approach was used to ensure denosumab has an effect greater than placebo (ie, the non-inferiority margin M1, ie, the lower bound of the two-sided 95% confidence interval 1.28, is ruled out). Next, a synthesis method was used for the non-inferiority test of the hypothesis that denosumab preserved at least 50% of the effect of zoledronic acid (HR [95% CI] of 1.48 [1.28, 1.71] for placebo vs zoledronic acid; p = 0.010, Cox proportional hazards model; Based on a Cox proportional hazards model stratified by the randomization stratification factors; Hazard Ratio (HR) = 0.98, 95% CI 2-sided [0.85 to 1.14] — A hazard ratio (denosumab:zoledronic acid) < 1 favors denosumab

2. Primary Outcome: Percentage of Participants With an On-study Skeletal Related Event
Description: A skeletal-related event (SRE) is defined as one of the following: pathologic fracture (vertebral or non-vertebral), radiation therapy to bone (including the use of radioisotopes), surgery to bone, or spinal cord compression.
Time Frame: as for outcome 1
Population: All randomized participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Zoledronic Acid | Denosumab
Number analyzed (Participants) | 859 | 859
percentage of participants | 44.6 [41.3 to 47.9] | 43.8 [40.5 to 47.1]

3. Primary Outcome: Kaplan-Meier Estimate of Percentage of Participants With an On-study Skeletal Related Event
Description: as for outcome 2
Time Frame: From randomization until the primary analysis data cut-off date of 19 July 2016 (per protocol); median time on study was 17.6 and 17.3 months in each treatment group respectively. The Kaplan-Meier estimate at weeks 25, 49 and 109 is reported.
Population: All randomized participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Zoledronic Acid | Denosumab
Number analyzed (Participants) | 859 | 859
percentage of participants
  At Week 25 | 36.5 [33.3 to 39.9] | 35.9 [32.7 to 39.3]
  At Week 49 | 43.2 [39.7 to 46.8] | 43.7 [40.2 to 47.3]
  At Week 109 | 50.6 [46.6 to 54.6] | 50.5 [46.6 to 54.5]

4. Secondary Outcome: Time to First On-study Skeletal Related Event - Superiority Analysis
Description: as for outcome 1
Time Frame: as for outcome 1
Population: All randomized participants
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Zoledronic Acid | Denosumab
Number analyzed (Participants) | 859 | 859
days | 730.0 [504.0 to 1014.0] | 695.0 [448.0 to NA] — Could not be estimated due to the low number of events
Statistical Analysis 1: Comparison: Zoledronic Acid vs Denosumab; Test type: Superiority — The statistical inferences of the treatment effect on secondary efficacy endpoints (time to the first on study SRE [superiority] and time to first and subsequent on study SRE [superiority, multiple event analysis]) were to be conducted if denosumab was determined to be non-inferior to zoledronic acid. To control the overall type I error for multiple comparisons at a significant level of 0.05, these secondary efficacy endpoints were tested simultaneously using the Hochberg procedure; p = 0.82, Log Rank; Based on a log rank test stratified by randomization stratification factors

5. Secondary Outcome: Time to First and Subsequent On-Study Skeletal Related Event - Number of Events Per Patient
Description: A skeletal-related event (SRE) is defined as one of the following: pathologic fracture (vertebral or non-vertebral), radiation therapy to bone (including the use of radioisotopes), surgery to bone, or spinal cord compression. Time to first on-study SRE is defined as the time interval (in days) from the randomization date to the date of first occurrence of on-study SRE. Time to a subsequent SRE is defined, similarly to the time to first on-study SRE, as the time interval from the randomization date to the date of a subsequent occurrence of on-study SRE, which had to be at least 21 days after the previous SRE.
  A multiple event analysis was used, which accounts for both the absolute number of SREs and for the time between two consecutive events, and therefore, provides a more sensitive assessment of the risk of experiencing an SRE. The average number of events per patient is reported.
Time Frame: as for outcome 1
Population: All randomized participants
Measure: Number; unit: events/patient
Arm/Group | Zoledronic Acid | Denosumab
Number analyzed (Participants) | 859 | 859
events/patient | 0.66 | 0.66
Statistical Analysis 1: Comparison: Zoledronic Acid vs Denosumab; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p = 0.84, Andersen-Gill model; Based on an Andersen-Gill model stratified by the randomization stratification factors; Rate ratio = 1.01, 95% CI 2-sided [0.89 to 1.15] — A rate ratio (denosumab:zoledronic acid) < 1 favors denosumab

6. Secondary Outcome: Time to First and Subsequent On-Study Skeletal Related Event - Number of Events
Description: A skeletal-related event (SRE) is defined as one of the following: pathologic fracture (vertebral or non-vertebral), radiation therapy to bone (including the use of radioisotopes), surgery to bone, or spinal cord compression. Time to first on-study SRE is defined as the time interval (in days) from the randomization date to the date of first occurrence of on-study SRE. Time to a subsequent SRE is defined, similarly to the time to first on-study SRE, as the time interval from the randomization date to the date of a subsequent occurrence of on-study SRE, which had to be at least 21 days after the previous SRE.
  A multiple event analysis was used, which accounts for both the absolute number of SREs and for the time between two consecutive events, and therefore, provides a more sensitive assessment of the risk of experiencing an SRE. The total number of events is reported.
Time Frame: as for outcome 1
Population: All randomized participants
Measure: Number; unit: skeletal-related events
Arm/Group | Zoledronic Acid | Denosumab
Number analyzed (Participants) | 859 | 859
skeletal-related events | 565 | 565

7. Secondary Outcome: Overall Survival
Description: Overall survival was defined as the time interval (in days) from the randomization date to the date of death. If a participant was still alive at the primary analysis data cut-off date or was lost to follow-up by the primary analysis data cut-off date, survival time was censored at their last contact date or the primary analysis data cut-off date, whichever was first.
Time Frame: as for outcome 1
Population: All randomized participants
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Zoledronic Acid | Denosumab
Number analyzed (Participants) | 859 | 859
days | NA [NA to NA] — Not estimable, the median survival and 95% CI were not reached | 1507.0 [NA to NA] — The 95% CI was not estimable as there were no participants in the risk set who survived at the median time
Statistical Analysis 1: Comparison: Zoledronic Acid vs Denosumab; The survival function of time to death for each treatment group was estimated using Kaplan-Meier method and the hazard ratio of denosumab compared with zoledronic acid and its 2-sided 95% CI were estimated using a Cox proportional hazards model stratified by the randomization stratification factors and including treatment groups, age, race group, geographic region, baseline creatinine clearance, baseline risk per cytogenetic based prognosis, and baseline ECOG as independent variables; Test type: Superiority — If superiority of denosumab over zoledronic acid was established for both time to first SRE and time to first and subsequent SRE, the additional secondary endpoint (overall survival) was to be tested at a significance level of 0.05; p = 0.41, Cox proportional hazards model; Hazard Ratio (HR) = 0.90, 95% CI 2-sided [0.70 to 1.16] — A hazard ratio (denosumab:zoledronic acid) < 1 favors denosumab

8. Secondary Outcome: Percentage of Participants Who Died
Time Frame: as for outcome 1
Population: All randomized participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Zoledronic Acid | Denosumab
Number analyzed (Participants) | 859 | 859
percentage of participants | 15.0 [12.6 to 17.4] | 14.1 [11.8 to 16.4]

ADVERSE EVENTS:
Time Frame: DB (double-blind treatment phase): adverse events (AEs) were from 1st dose of study drug to the later of 30 days after last dose or end of treatment phase. OL (open-label treatment phase): AEs were from 1st dose of OL study drug to end of study. Median months on study drug: 18.4 (zoledronic acid [ZA]) and 19.4 (Denosumab [Dmab]) in DB; 23.2 (ZA/Dmab) and 23.0 (Dmab/Dmab) in OL.
Groups:
- DB: Zoledronic Acid: Participants received zoledronic acid 4 mg intravenously plus placebo to denosumab subcutaneously once every 4 weeks (Q4W) in the double-blind (DB) treatment phase.
- DB: Denosumab: Participants received denosumab 120 mg subcutaneously plus placebo to zoledronic acid intravenously once every 4 weeks (Q4W) in the double-blind (DB) treatment phase.
- OL: Zoledronic Acid / Denosumab: Participants who received zoledronic acid 4 mg intravenously plus placebo to denosumab subcutaneously (SC) once every 4 weeks (Q4W) in the double-blind treatment phase received denosumab 120 mg SC Q4W in the open-label (OL) treatment phase.
- OL: Denosumab / Denosumab: Participants who received denosumab 120 mg subcutaneously (SC) plus placebo to zoledronic acid intravenously once every 4 weeks (Q4W) in the double-blind treatment phase received denosumab 120 mg SC Q4W in the open-label (OL) treatment phase.
Arm/Group | DB: Zoledronic Acid | DB: Denosumab | OL: Zoledronic Acid / Denosumab | OL: Denosumab / Denosumab
Serious Adverse Events (participants affected / at risk) | 447/852 | 434/850 | 159/418 | 156/426
Other Adverse Events (participants affected / at risk) | 778/852 | 757/850 | 313/418 | 312/426
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DB: Zoledronic Acid (N=852) | DB: Denosumab (N=850) | OL: Zoledronic Acid / Denosumab (N=418) | OL: Denosumab / Denosumab (N=426)
Agranulocytosis (Blood and lymphatic system disorders) | 1 | 1 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 26 | 12 | 5 | 8
Autoimmune haemolytic anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Bicytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Bone marrow failure (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 25 | 23 | 7 | 6
Haemolytic anaemia (Blood and lymphatic system disorders) | 1 | 1 | 0 | 0
Hyperviscosity syndrome (Blood and lymphatic system disorders) | 0 | 3 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 2 | 2 | 2 | 1
Neutropenia (Blood and lymphatic system disorders) | 13 | 4 | 4 | 3
Pancytopenia (Blood and lymphatic system disorders) | 4 | 2 | 3 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 12 | 9 | 2 | 7
Acute coronary syndrome (Cardiac disorders) | 1 | 2 | 3 | 0
Acute myocardial infarction (Cardiac disorders) | 6 | 2 | 1 | 1
Angina pectoris (Cardiac disorders) | 2 | 2 | 1 | 0
Angina unstable (Cardiac disorders) | 1 | 0 | 2 | 0
Atrial fibrillation (Cardiac disorders) | 10 | 4 | 2 | 1
Atrial flutter (Cardiac disorders) | 0 | 1 | 1 | 0
Atrial tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0
Bradycardia (Cardiac disorders) | 4 | 0 | 0 | 0
Cardiac amyloidosis (Cardiac disorders) | 1 | 0 | 1 | 0
Cardiac arrest (Cardiac disorders) | 11 | 6 | 1 | 1
Cardiac disorder (Cardiac disorders) | 0 | 1 | 0 | 0
Cardiac failure (Cardiac disorders) | 7 | 11 | 3 | 4
Cardiac failure acute (Cardiac disorders) | 2 | 1 | 0 | 0
Cardiac failure chronic (Cardiac disorders) | 0 | 3 | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 5 | 5 | 1 | 3
Cardio-respiratory arrest (Cardiac disorders) | 2 | 0 | 1 | 0
Cardiopulmonary failure (Cardiac disorders) | 2 | 0 | 0 | 0
Cardiovascular insufficiency (Cardiac disorders) | 1 | 1 | 0 | 0
Coronary artery disease (Cardiac disorders) | 1 | 2 | 0 | 0
Left ventricular failure (Cardiac disorders) | 0 | 1 | 0 | 1
Mitral valve stenosis (Cardiac disorders) | 0 | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 2 | 1 | 0 | 2
Myocardial ischaemia (Cardiac disorders) | 1 | 2 | 0 | 1
Myocarditis (Cardiac disorders) | 1 | 2 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 1 | 0 | 1
Pericarditis (Cardiac disorders) | 0 | 1 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 1 | 0 | 0 | 0
Sinus node dysfunction (Cardiac disorders) | 1 | 0 | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 2 | 3 | 0 | 1
Tachyarrhythmia (Cardiac disorders) | 0 | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0
Tricuspid valve incompetence (Cardiac disorders) | 0 | 1 | 0 | 0
Aplasia (Congenital, familial and genetic disorders) | 0 | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 1 | 0 | 0
Vertigo positional (Ear and labyrinth disorders) | 1 | 1 | 0 | 0
Adrenal insufficiency (Endocrine disorders) | 0 | 1 | 0 | 0
Hypercalcaemia of malignancy (Endocrine disorders) | 1 | 0 | 0 | 0
Hyperparathyroidism primary (Endocrine disorders) | 1 | 0 | 0 | 0
Steroid withdrawal syndrome (Endocrine disorders) | 1 | 0 | 0 | 0
Cataract (Eye disorders) | 2 | 0 | 2 | 0
Diplopia (Eye disorders) | 1 | 1 | 0 | 0
Exophthalmos (Eye disorders) | 1 | 0 | 0 | 0
Extraocular muscle paresis (Eye disorders) | 1 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Abdominal hernia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Abdominal incarcerated hernia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 5 | 1 | 4 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 2 | 2 | 0 | 0
Abdominal wall haematoma (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Chronic gastritis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 1 | 2 | 1 | 1
Colitis ischaemic (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 4 | 3 | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 10 | 9 | 1 | 4
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Diverticulum intestinal (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Duodenal ulcer (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 3 | 0 | 1
Enteritis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 1 | 2 | 0 | 0
Gastritis erosive (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastrointestinal amyloidosis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 5 | 3 | 1 | 1
Gastrointestinal perforation (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Gingivitis ulcerative (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Hiatus hernia (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Inguinal hernia (Gastrointestinal disorders) | 2 | 2 | 1 | 3
Intestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 3 | 1 | 2 | 0
Large intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Large intestine perforation (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Large intestine polyp (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 0 | 0 | 2
Mechanical ileus (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Melaena (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Mouth haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 4 | 4 | 1 | 0
Oesophagitis (Gastrointestinal disorders) | 2 | 1 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Proctitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 4 | 1 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Subileus (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Umbilical hernia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 11 | 7 | 3 | 3
Asthenia (General disorders) | 7 | 3 | 1 | 5
Chest pain (General disorders) | 0 | 1 | 0 | 0
Chills (General disorders) | 1 | 1 | 0 | 0
Death (General disorders) | 3 | 3 | 1 | 1
Disease progression (General disorders) | 1 | 2 | 0 | 0
Fatigue (General disorders) | 1 | 1 | 2 | 0
Gait disturbance (General disorders) | 1 | 2 | 0 | 0
General physical health deterioration (General disorders) | 10 | 10 | 2 | 6
Generalised oedema (General disorders) | 0 | 3 | 0 | 0
Hyperpyrexia (General disorders) | 1 | 1 | 0 | 0
Hyperthermia (General disorders) | 1 | 0 | 1 | 0
Localised oedema (General disorders) | 0 | 1 | 0 | 0
Malaise (General disorders) | 0 | 2 | 0 | 0
Mucosal ulceration (General disorders) | 0 | 1 | 0 | 0
Multiple organ dysfunction syndrome (General disorders) | 6 | 5 | 3 | 1
Non-cardiac chest pain (General disorders) | 5 | 4 | 0 | 2
Oedema peripheral (General disorders) | 3 | 5 | 2 | 1
Performance status decreased (General disorders) | 0 | 1 | 1 | 0
Pyrexia (General disorders) | 28 | 24 | 2 | 4
Sudden cardiac death (General disorders) | 1 | 1 | 0 | 0
Sudden death (General disorders) | 5 | 3 | 1 | 1
Acute hepatic failure (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Bile duct stenosis (Hepatobiliary disorders) | 0 | 1 | 1 | 0
Cholangitis acute (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 2 | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 2 | 0 | 2 | 1
Drug-induced liver injury (Hepatobiliary disorders) | 1 | 2 | 0 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 2 | 0 | 0
Hepatitis toxic (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Acute graft versus host disease (Immune system disorders) | 0 | 1 | 0 | 0
Acute graft versus host disease in intestine (Immune system disorders) | 0 | 1 | 0 | 0
Anaphylactic reaction (Immune system disorders) | 1 | 1 | 0 | 0
Hypersensitivity (Immune system disorders) | 1 | 0 | 0 | 0
Abscess bacterial (Infections and infestations) | 0 | 1 | 0 | 0
Adenoviral haemorrhagic cystitis (Infections and infestations) | 1 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 3 | 2 | 1 | 1
Arthritis bacterial (Infections and infestations) | 1 | 1 | 0 | 0
Arthritis infective (Infections and infestations) | 0 | 1 | 1 | 0
Atypical pneumonia (Infections and infestations) | 1 | 0 | 0 | 0
Bacteraemia (Infections and infestations) | 2 | 1 | 1 | 0
Bacterial infection (Infections and infestations) | 1 | 3 | 0 | 0
Bacterial pyelonephritis (Infections and infestations) | 0 | 1 | 0 | 1
Bacterial sepsis (Infections and infestations) | 0 | 1 | 0 | 0
Bronchiolitis (Infections and infestations) | 2 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 7 | 11 | 4 | 2
Bursitis infective (Infections and infestations) | 0 | 1 | 0 | 0
Cellulitis (Infections and infestations) | 5 | 4 | 0 | 4
Cellulitis orbital (Infections and infestations) | 0 | 1 | 0 | 0
Cholecystitis infective (Infections and infestations) | 0 | 1 | 0 | 0
Chronic sinusitis (Infections and infestations) | 0 | 1 | 0 | 0
Clostridium bacteraemia (Infections and infestations) | 0 | 1 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 4 | 6 | 1 | 2
Clostridium difficile infection (Infections and infestations) | 0 | 3 | 1 | 1
Creutzfeldt-Jakob disease (Infections and infestations) | 0 | 1 | 0 | 0
Cystitis (Infections and infestations) | 1 | 0 | 0 | 0
Cytomegalovirus chorioretinitis (Infections and infestations) | 1 | 0 | 0 | 0
Cytomegalovirus infection (Infections and infestations) | 1 | 2 | 0 | 0
Device related infection (Infections and infestations) | 2 | 3 | 1 | 1
Diarrhoea infectious (Infections and infestations) | 1 | 0 | 0 | 0
Diverticulitis (Infections and infestations) | 1 | 3 | 1 | 1
Encephalitis (Infections and infestations) | 1 | 0 | 0 | 0
Erysipelas (Infections and infestations) | 2 | 1 | 0 | 0
Escherichia sepsis (Infections and infestations) | 1 | 0 | 0 | 0
Escherichia urinary tract infection (Infections and infestations) | 1 | 1 | 0 | 0
Extradural abscess (Infections and infestations) | 1 | 0 | 0 | 0
Febrile infection (Infections and infestations) | 2 | 2 | 0 | 0
Folliculitis (Infections and infestations) | 1 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 3 | 1 | 1 | 2
Gastroenteritis viral (Infections and infestations) | 0 | 2 | 0 | 1
Gingivitis (Infections and infestations) | 1 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 9 | 5 | 1 | 0
Human herpesvirus 6 infection (Infections and infestations) | 1 | 0 | 0 | 0
Infection (Infections and infestations) | 0 | 3 | 0 | 0
Infection in an immunocompromised host (Infections and infestations) | 1 | 0 | 0 | 0
Infection reactivation (Infections and infestations) | 0 | 1 | 0 | 0
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 0 | 1 | 0 | 0
Influenza (Infections and infestations) | 6 | 10 | 3 | 5
Intervertebral discitis (Infections and infestations) | 1 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 12 | 5 | 0 | 1
Lower respiratory tract infection fungal (Infections and infestations) | 1 | 1 | 0 | 0
Lower respiratory tract infection viral (Infections and infestations) | 1 | 0 | 0 | 0
Lung infection (Infections and infestations) | 0 | 2 | 2 | 1
Meningitis meningococcal (Infections and infestations) | 0 | 1 | 0 | 0
Meningitis pneumococcal (Infections and infestations) | 0 | 1 | 0 | 0
Necrotising fasciitis (Infections and infestations) | 0 | 1 | 0 | 0
Neutropenic infection (Infections and infestations) | 1 | 0 | 0 | 0
Neutropenic sepsis (Infections and infestations) | 3 | 2 | 0 | 0
Osteomyelitis (Infections and infestations) | 1 | 3 | 1 | 0
Otitis media (Infections and infestations) | 1 | 0 | 0 | 0
Parainfluenzae virus infection (Infections and infestations) | 3 | 0 | 0 | 0
Perineal abscess (Infections and infestations) | 0 | 1 | 0 | 0
Periodontitis (Infections and infestations) | 1 | 0 | 0 | 0
Peritonitis (Infections and infestations) | 0 | 2 | 1 | 0
Peritonsillar abscess (Infections and infestations) | 0 | 1 | 0 | 0
Pneumococcal sepsis (Infections and infestations) | 1 | 1 | 0 | 0
Pneumocystis jirovecii infection (Infections and infestations) | 1 | 0 | 0 | 0
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 82 | 79 | 34 | 31
Pneumonia bacterial (Infections and infestations) | 0 | 2 | 0 | 1
Pneumonia klebsiella (Infections and infestations) | 0 | 1 | 0 | 0
Pneumonia legionella (Infections and infestations) | 1 | 1 | 0 | 0
Pneumonia pneumococcal (Infections and infestations) | 0 | 1 | 0 | 0
Pneumonia respiratory syncytial viral (Infections and infestations) | 0 | 1 | 0 | 0
Pneumonia staphylococcal (Infections and infestations) | 1 | 1 | 0 | 0
Pneumonia viral (Infections and infestations) | 1 | 1 | 1 | 1
Post procedural infection (Infections and infestations) | 1 | 0 | 0 | 0
Post procedural sepsis (Infections and infestations) | 0 | 1 | 0 | 0
Postoperative wound infection (Infections and infestations) | 1 | 0 | 1 | 0
Pseudomonal sepsis (Infections and infestations) | 1 | 0 | 0 | 0
Pulmonary mycosis (Infections and infestations) | 0 | 1 | 0 | 0
Respiratory tract infection (Infections and infestations) | 8 | 7 | 8 | 5
Respiratory tract infection fungal (Infections and infestations) | 1 | 0 | 0 | 0
Respiratory tract infection viral (Infections and infestations) | 1 | 0 | 0 | 1
Salmonellosis (Infections and infestations) | 1 | 1 | 0 | 0
Scrotal abscess (Infections and infestations) | 0 | 1 | 0 | 0
Sepsis (Infections and infestations) | 24 | 19 | 8 | 11
Sepsis syndrome (Infections and infestations) | 0 | 1 | 1 | 0
Septic necrosis (Infections and infestations) | 0 | 1 | 0 | 0
Septic shock (Infections and infestations) | 7 | 6 | 7 | 2
Sinusitis (Infections and infestations) | 2 | 2 | 0 | 1
Spinal cord infection (Infections and infestations) | 1 | 0 | 1 | 0
Staphylococcal bacteraemia (Infections and infestations) | 2 | 0 | 0 | 0
Staphylococcal sepsis (Infections and infestations) | 2 | 1 | 0 | 0
Staphylococcal skin infection (Infections and infestations) | 1 | 0 | 0 | 0
Tonsillitis (Infections and infestations) | 1 | 0 | 0 | 0
Tracheobronchitis (Infections and infestations) | 0 | 2 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 7 | 2 | 2
Urinary tract infection (Infections and infestations) | 9 | 6 | 2 | 1
Urinary tract infection bacterial (Infections and infestations) | 1 | 0 | 1 | 0
Urosepsis (Infections and infestations) | 1 | 3 | 0 | 1
Varicella (Infections and infestations) | 0 | 1 | 0 | 0
Viral infection (Infections and infestations) | 3 | 2 | 1 | 0
Viral myositis (Infections and infestations) | 1 | 0 | 0 | 0
Wound infection (Infections and infestations) | 1 | 0 | 0 | 0
Abdominal injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Anastomotic leak (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Bone contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Brain contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0
Concussion (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 6 | 3 | 0 | 3
Femoral neck fracture (Injury, poisoning and procedural complications) | 7 | 2 | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Hand fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 2 | 3 | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 2 | 1 | 0 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 8 | 4 | 0 | 1
Patella fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 2 | 1 | 0 | 2
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 3
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Sternal fracture (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 5 | 6 | 0 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Transfusion related complication (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 3 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 3 | 1 | 0
Bilirubin conjugated increased (Investigations) | 0 | 1 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 1 | 0 | 0
Blood creatine increased (Investigations) | 0 | 1 | 0 | 0
Blood creatinine increased (Investigations) | 3 | 2 | 1 | 1
Blood electrolytes abnormal (Investigations) | 1 | 0 | 0 | 0
Blood immunoglobulin G increased (Investigations) | 1 | 0 | 0 | 0
Blood immunoglobulin M increased (Investigations) | 2 | 1 | 0 | 0
Blood lactate dehydrogenase increased (Investigations) | 1 | 0 | 0 | 0
Body temperature increased (Investigations) | 1 | 0 | 0 | 0
Bone marrow plasmacyte count increased (Investigations) | 2 | 1 | 0 | 0
C-reactive protein increased (Investigations) | 0 | 1 | 0 | 0
Chest X-ray abnormal (Investigations) | 1 | 0 | 0 | 0
Eastern Cooperative Oncology Group performance status worsened (Investigations) | 0 | 1 | 0 | 0
Haemoglobin decreased (Investigations) | 1 | 1 | 0 | 1
Heart rate irregular (Investigations) | 0 | 1 | 0 | 0
Light chain analysis increased (Investigations) | 1 | 0 | 0 | 0
Liver function test abnormal (Investigations) | 1 | 1 | 0 | 0
Monoclonal immunoglobulin present (Investigations) | 1 | 2 | 1 | 1
Neutrophil count decreased (Investigations) | 0 | 1 | 0 | 1
Platelet count decreased (Investigations) | 6 | 2 | 1 | 2
Weight decreased (Investigations) | 1 | 1 | 0 | 0
White blood cell count decreased (Investigations) | 0 | 1 | 0 | 1
Cachexia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 2 | 2 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 12 | 10 | 3 | 1
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 | 2 | 0 | 0
Failure to thrive (Metabolism and nutrition disorders) | 3 | 1 | 1 | 1
Fluid imbalance (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Gout (Metabolism and nutrition disorders) | 2 | 2 | 0 | 0
Haemosiderosis (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 8 | 2 | 0 | 3
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 3 | 1 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hyperproteinaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 2 | 8 | 2 | 2
Hypoglycaemia (Metabolism and nutrition disorders) | 2 | 3 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 7 | 1 | 0 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 3 | 3 | 0 | 0
Lactic acidosis (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Tumour lysis syndrome (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 3 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 16 | 9 | 1 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 7 | 1 | 3 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 0
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 3 | 3 | 1 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 | 2 | 0 | 0
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 2 | 2 | 0 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 13 | 18 | 11 | 12
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 | 3 | 1 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 1
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Vertebral lesion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 1 | 0
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 3 | 1
Basosquamous carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0 | 0
Bladder cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Chronic myelomonocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 3 | 1 | 0
Colorectal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Malignant neoplasm of pleura (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Malignant neoplasm of renal pelvis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 1 | 0
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0
Neoplasm of orbit (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Neuroendocrine tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Non-small cell lung cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Paraproteinaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 3 | 0 | 0
Plasma cell leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 1 | 1 | 2
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 16 | 18 | 3 | 10
Plasma cell myeloma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Plasmacytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 7 | 1 | 5
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 3 | 1 | 1
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0 | 1 | 0
Basilar migraine (Nervous system disorders) | 0 | 1 | 0 | 0
Brain injury (Nervous system disorders) | 1 | 0 | 0 | 0
Cauda equina syndrome (Nervous system disorders) | 1 | 0 | 0 | 0
Cerebral haemorrhage (Nervous system disorders) | 4 | 0 | 2 | 1
Cerebral ischaemia (Nervous system disorders) | 3 | 2 | 1 | 0
Cerebral vasoconstriction (Nervous system disorders) | 0 | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 5 | 5 | 0 | 1
Cognitive disorder (Nervous system disorders) | 0 | 1 | 0 | 0
Coma (Nervous system disorders) | 1 | 0 | 0 | 0
Depressed level of consciousness (Nervous system disorders) | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 4 | 2 | 0 | 0
Encephalopathy (Nervous system disorders) | 3 | 2 | 2 | 0
Epilepsy (Nervous system disorders) | 0 | 1 | 0 | 0
Generalised tonic-clonic seizure (Nervous system disorders) | 0 | 1 | 0 | 0
Haemorrhage intracranial (Nervous system disorders) | 3 | 1 | 0 | 0
Haemorrhagic stroke (Nervous system disorders) | 0 | 1 | 0 | 0
Hemiparesis (Nervous system disorders) | 1 | 1 | 0 | 0
Hemiplegia (Nervous system disorders) | 1 | 0 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 0 | 1 | 0
Ischaemic cerebral infarction (Nervous system disorders) | 1 | 0 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 1 | 3 | 1 | 1
Lacunar infarction (Nervous system disorders) | 0 | 2 | 0 | 0
Loss of consciousness (Nervous system disorders) | 2 | 0 | 0 | 0
Lumbosacral radiculopathy (Nervous system disorders) | 0 | 1 | 0 | 0
Nerve degeneration (Nervous system disorders) | 0 | 1 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 1 | 1 | 0 | 0
Paralysis (Nervous system disorders) | 1 | 0 | 0 | 0
Paraparesis (Nervous system disorders) | 2 | 0 | 0 | 0
Paraplegia (Nervous system disorders) | 0 | 1 | 0 | 0
Paresis (Nervous system disorders) | 0 | 1 | 0 | 0
Polyneuropathy (Nervous system disorders) | 1 | 1 | 0 | 0
Presyncope (Nervous system disorders) | 1 | 0 | 1 | 0
Radiculopathy (Nervous system disorders) | 2 | 0 | 0 | 0
Sciatica (Nervous system disorders) | 2 | 2 | 0 | 0
Seizure (Nervous system disorders) | 1 | 3 | 0 | 1
Seizure like phenomena (Nervous system disorders) | 0 | 1 | 0 | 0
Spinal cord compression (Nervous system disorders) | 8 | 4 | 0 | 1
Subarachnoid haemorrhage (Nervous system disorders) | 1 | 1 | 1 | 0
Syncope (Nervous system disorders) | 9 | 7 | 0 | 2
Transient ischaemic attack (Nervous system disorders) | 1 | 1 | 0 | 1
Device breakage (Product Issues) | 1 | 0 | 0 | 0
Device failure (Product Issues) | 0 | 1 | 0 | 0
Device occlusion (Product Issues) | 0 | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 1 | 0 | 0
Completed suicide (Psychiatric disorders) | 2 | 0 | 1 | 0
Confusional state (Psychiatric disorders) | 3 | 5 | 0 | 0
Delirium (Psychiatric disorders) | 2 | 4 | 0 | 2
Depression (Psychiatric disorders) | 0 | 3 | 0 | 1
Disorientation (Psychiatric disorders) | 0 | 1 | 0 | 0
Major depression (Psychiatric disorders) | 1 | 0 | 0 | 0
Mental status changes (Psychiatric disorders) | 0 | 1 | 0 | 1
Mutism (Psychiatric disorders) | 1 | 0 | 0 | 0
Psychotic disorder (Psychiatric disorders) | 0 | 1 | 0 | 0
Suicide attempt (Psychiatric disorders) | 1 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 24 | 17 | 8 | 2
Bladder perforation (Renal and urinary disorders) | 0 | 1 | 0 | 0
Chronic kidney disease (Renal and urinary disorders) | 1 | 2 | 0 | 1
Cystitis haemorrhagic (Renal and urinary disorders) | 0 | 1 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 1 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 0 | 0
Renal colic (Renal and urinary disorders) | 0 | 2 | 1 | 0
Renal disorder (Renal and urinary disorders) | 0 | 1 | 0 | 0
Renal failure (Renal and urinary disorders) | 7 | 4 | 1 | 6
Renal impairment (Renal and urinary disorders) | 1 | 2 | 1 | 1
Ureteric obstruction (Renal and urinary disorders) | 0 | 1 | 0 | 0
Ureterolithiasis (Renal and urinary disorders) | 0 | 1 | 0 | 0
Urinary retention (Renal and urinary disorders) | 2 | 2 | 2 | 0
Adenomyosis (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 1 | 0 | 1
Scrotal oedema (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Testicular mass (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 2 | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Bronchopneumopathy (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 4 | 4 | 3 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 10 | 5 | 2 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 0 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 1 | 1
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Non-cardiogenic pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 | 6 | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 6 | 2 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Pulmonary artery thrombosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 13 | 16 | 5 | 3
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 2 | 3
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 11 | 4 | 4 | 2
Stridor (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 2 | 0 | 1 | 0
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0
Keloid scar (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Purpura (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Skin disorder (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Cataract operation (Surgical and medical procedures) | 1 | 0 | 0 | 0
Fistula repair (Surgical and medical procedures) | 1 | 0 | 0 | 0
Haematopoietic stem cell mobilisation (Surgical and medical procedures) | 0 | 2 | 0 | 0
Internal fixation of fracture (Surgical and medical procedures) | 0 | 1 | 0 | 0
Intra-uterine contraceptive device removal (Surgical and medical procedures) | 0 | 1 | 0 | 0
Knee arthroplasty (Surgical and medical procedures) | 1 | 0 | 0 | 0
Rehabilitation therapy (Surgical and medical procedures) | 0 | 1 | 0 | 0
Aortic aneurysm (Vascular disorders) | 1 | 0 | 0 | 0
Aortic aneurysm rupture (Vascular disorders) | 1 | 0 | 0 | 0
Aortic dissection (Vascular disorders) | 1 | 1 | 0 | 0
Aortic dissection rupture (Vascular disorders) | 1 | 0 | 0 | 0
Aortic thrombosis (Vascular disorders) | 0 | 1 | 0 | 0
Circulatory collapse (Vascular disorders) | 4 | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 8 | 11 | 2 | 1
Essential hypertension (Vascular disorders) | 1 | 0 | 0 | 0
Haematoma (Vascular disorders) | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 4 | 0 | 1
Hypotension (Vascular disorders) | 1 | 2 | 1 | 0
Hypovolaemic shock (Vascular disorders) | 0 | 1 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 3 | 1 | 0 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 1 | 0 | 0
Peripheral artery aneurysm (Vascular disorders) | 0 | 1 | 0 | 0
Peripheral ischaemia (Vascular disorders) | 0 | 1 | 2 | 0
Superior vena cava syndrome (Vascular disorders) | 0 | 1 | 0 | 0
Thrombophlebitis superficial (Vascular disorders) | 1 | 1 | 0 | 0
Thrombosis (Vascular disorders) | 0 | 1 | 0 | 1
Vasospasm (Vascular disorders) | 1 | 0 | 0 | 0
Acquired haemophilia with anti FVIII, XI, or XIII (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Anaemia of malignant disease (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Cytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1
Platelet disorder (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Thrombocytosis (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Acute left ventricular failure (Cardiac disorders) | 0 | 0 | 1 | 0
Arrhythmia (Cardiac disorders) | 0 | 0 | 0 | 1
Cardiac tamponade (Cardiac disorders) | 0 | 0 | 1 | 0
Cardiac valve disease (Cardiac disorders) | 0 | 1 | 0 | 0
Cardiomyopathy (Cardiac disorders) | 0 | 1 | 0 | 0
Left ventricular dysfunction (Cardiac disorders) | 1 | 0 | 0 | 0
Pericardial effusion (Cardiac disorders) | 0 | 1 | 0 | 0
Ventricular arrhythmia (Cardiac disorders) | 1 | 0 | 0 | 0
Odontogenic cyst (Congenital, familial and genetic disorders) | 0 | 1 | 0 | 0
Adrenocortical insufficiency acute (Endocrine disorders) | 0 | 1 | 0 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 1 | 0 | 0
Ulcerative keratitis (Eye disorders) | 0 | 0 | 0 | 1
Vision blurred (Eye disorders) | 0 | 1 | 0 | 0
Anal fissure (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Appendiceal mucocoele (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Crohn's disease (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Gastrointestinal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gingival bleeding (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Intestinal ischaemia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Jejunal perforation (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Large intestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Obstructive pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Retroperitoneal mass (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Small intestinal perforation (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Toothache (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Oedema (General disorders) | 0 | 0 | 0 | 2
Systemic inflammatory response syndrome (General disorders) | 0 | 0 | 0 | 1
Bile duct obstruction (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Cholecystitis chronic (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Gallbladder rupture (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Hepatic failure (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Hepatitis (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Hepatotoxicity (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Jaundice cholestatic (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Serum sickness (Immune system disorders) | 0 | 0 | 1 | 0
Abdominal abscess (Infections and infestations) | 0 | 1 | 0 | 0
Abscess jaw (Infections and infestations) | 0 | 1 | 0 | 0
Abscess neck (Infections and infestations) | 1 | 0 | 0 | 0
Abscess soft tissue (Infections and infestations) | 0 | 0 | 2 | 0
Acute sinusitis (Infections and infestations) | 0 | 1 | 0 | 0
Bacterial parotitis (Infections and infestations) | 0 | 1 | 0 | 0
Bronchopulmonary aspergillosis (Infections and infestations) | 0 | 0 | 2 | 0
Campylobacter gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 1
Candida infection (Infections and infestations) | 0 | 0 | 1 | 0
Device related sepsis (Infections and infestations) | 1 | 0 | 0 | 0
Empyema (Infections and infestations) | 0 | 0 | 1 | 0
Endocarditis (Infections and infestations) | 0 | 0 | 1 | 0
Enterocolitis bacterial (Infections and infestations) | 0 | 0 | 1 | 0
Epiglottitis (Infections and infestations) | 1 | 0 | 0 | 0
Gangrene (Infections and infestations) | 0 | 0 | 1 | 0
Gastroenteritis norovirus (Infections and infestations) | 1 | 0 | 0 | 0
Gastroenteritis salmonella (Infections and infestations) | 0 | 1 | 0 | 0
Gastrointestinal infection (Infections and infestations) | 0 | 0 | 1 | 0
Hepatitis B (Infections and infestations) | 0 | 0 | 1 | 0
Herpes virus infection (Infections and infestations) | 1 | 0 | 0 | 0
Herpes zoster cutaneous disseminated (Infections and infestations) | 0 | 0 | 0 | 1
Infected dermal cyst (Infections and infestations) | 0 | 0 | 1 | 0
Large intestine infection (Infections and infestations) | 1 | 1 | 0 | 0
Meningitis (Infections and infestations) | 1 | 0 | 0 | 0
Meningitis cryptococcal (Infections and infestations) | 0 | 0 | 1 | 0
Metapneumovirus infection (Infections and infestations) | 0 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 1 | 0
Opportunistic infection (Infections and infestations) | 0 | 0 | 1 | 0
Otitis externa (Infections and infestations) | 0 | 0 | 0 | 1
Parvovirus B19 infection (Infections and infestations) | 0 | 0 | 0 | 1
Pleural infection (Infections and infestations) | 0 | 0 | 1 | 0
Pneumonia fungal (Infections and infestations) | 0 | 0 | 0 | 1
Pneumonia haemophilus (Infections and infestations) | 0 | 0 | 1 | 0
Pneumonia pseudomonal (Infections and infestations) | 0 | 0 | 1 | 0
Pneumonia streptococcal (Infections and infestations) | 0 | 0 | 0 | 1
Pseudomembranous colitis (Infections and infestations) | 0 | 0 | 1 | 0
Pulmonary sepsis (Infections and infestations) | 1 | 0 | 0 | 0
Soft tissue infection (Infections and infestations) | 0 | 1 | 0 | 0
Urinary tract infection fungal (Infections and infestations) | 0 | 0 | 1 | 0
Vascular device infection (Infections and infestations) | 0 | 1 | 0 | 1
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Compression fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Incarcerated incisional hernia (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Poisoning (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0
Post procedural fever (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Procedural nausea (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Pulmonary contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Blood immunoglobulin A increased (Investigations) | 1 | 1 | 0 | 0
Influenza A virus test positive (Investigations) | 0 | 1 | 0 | 1
Light chain analysis abnormal (Investigations) | 0 | 0 | 1 | 0
Plasma cells increased (Investigations) | 0 | 0 | 1 | 0
Plasma cells present (Investigations) | 0 | 0 | 0 | 1
Protein urine present (Investigations) | 0 | 0 | 1 | 1
White blood cell count increased (Investigations) | 0 | 0 | 0 | 1
Hyperglycaemic hyperosmolar nonketotic syndrome (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Obesity (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Steroid diabetes (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Bone lesion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Bone swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Mobility decreased (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Osteolysis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Acute leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 2
Acute lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Acute lymphocytic leukaemia recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Anaplastic large-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Bone marrow tumour cell infiltration (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Glioblastoma multiforme (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0 | 0
Oropharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Spinal cord neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Brain oedema (Nervous system disorders) | 0 | 0 | 1 | 0
Cerebral atrophy (Nervous system disorders) | 0 | 1 | 0 | 0
Cerebral haematoma (Nervous system disorders) | 0 | 1 | 0 | 0
Cerebral infarction (Nervous system disorders) | 1 | 0 | 0 | 0
Cerebrovascular disorder (Nervous system disorders) | 0 | 0 | 0 | 1
Cervical cord compression (Nervous system disorders) | 0 | 1 | 0 | 0
Dementia (Nervous system disorders) | 0 | 0 | 1 | 0
Encephalitis post varicella (Nervous system disorders) | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 0 | 1
Intracranial mass (Nervous system disorders) | 0 | 1 | 0 | 0
Myelopathy (Nervous system disorders) | 0 | 1 | 0 | 0
Parkinson's disease (Nervous system disorders) | 0 | 0 | 1 | 0
Device dislocation (Product Issues) | 1 | 0 | 0 | 0
Adjustment disorder (Psychiatric disorders) | 0 | 0 | 0 | 1
Drug dependence (Psychiatric disorders) | 1 | 0 | 0 | 1
Organic brain syndrome (Psychiatric disorders) | 0 | 1 | 0 | 0
Psychiatric decompensation (Psychiatric disorders) | 0 | 0 | 0 | 1
Bladder obstruction (Renal and urinary disorders) | 1 | 0 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 0 | 1
Nephropathy toxic (Renal and urinary disorders) | 0 | 0 | 1 | 0
Oliguria (Renal and urinary disorders) | 0 | 0 | 1 | 0
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Pleural disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pleural thickening (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0
Rash generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Autologous haematopoietic stem cell transplant (Surgical and medical procedures) | 0 | 2 | 0 | 0
Aortic stenosis (Vascular disorders) | 0 | 0 | 1 | 1
Arterial disorder (Vascular disorders) | 1 | 0 | 0 | 0
Hypertensive urgency (Vascular disorders) | 0 | 1 | 0 | 1
Venous thrombosis (Vascular disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | DB: Zoledronic Acid (N=852) | DB: Denosumab (N=850) | OL: Zoledronic Acid / Denosumab (N=418) | OL: Denosumab / Denosumab (N=426)
Anaemia (Blood and lymphatic system disorders) | 185 | 208 | 51 | 62
Febrile neutropenia (Blood and lymphatic system disorders) | 82 | 89 | 9 | 2
Neutropenia (Blood and lymphatic system disorders) | 166 | 173 | 40 | 51
Thrombocytopenia (Blood and lymphatic system disorders) | 151 | 174 | 27 | 27
Abdominal pain (Gastrointestinal disorders) | 49 | 78 | 16 | 13
Constipation (Gastrointestinal disorders) | 214 | 207 | 19 | 27
Diarrhoea (Gastrointestinal disorders) | 301 | 304 | 73 | 57
Dyspepsia (Gastrointestinal disorders) | 62 | 60 | 12 | 11
Nausea (Gastrointestinal disorders) | 274 | 284 | 32 | 35
Stomatitis (Gastrointestinal disorders) | 53 | 63 | 5 | 8
Vomiting (Gastrointestinal disorders) | 159 | 147 | 18 | 19
Asthenia (General disorders) | 128 | 112 | 26 | 18
Fatigue (General disorders) | 215 | 206 | 43 | 38
Mucosal inflammation (General disorders) | 55 | 76 | 5 | 3
Oedema peripheral (General disorders) | 147 | 152 | 29 | 14
Pyrexia (General disorders) | 210 | 182 | 30 | 44
Bronchitis (Infections and infestations) | 72 | 72 | 31 | 32
Herpes zoster (Infections and infestations) | 68 | 62 | 13 | 5
Nasopharyngitis (Infections and infestations) | 79 | 84 | 42 | 38
Respiratory tract infection (Infections and infestations) | 53 | 56 | 25 | 26
Upper respiratory tract infection (Infections and infestations) | 127 | 143 | 62 | 58
Urinary tract infection (Infections and infestations) | 51 | 63 | 17 | 19
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 72 | 70 | 1 | 1
Rib fracture (Injury, poisoning and procedural complications) | 70 | 69 | 2 | 3
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 75 | 95 | 0 | 1
Blood creatinine increased (Investigations) | 80 | 36 | 15 | 9
Platelet count decreased (Investigations) | 55 | 55 | 10 | 14
Weight decreased (Investigations) | 61 | 61 | 12 | 9
Decreased appetite (Metabolism and nutrition disorders) | 166 | 140 | 12 | 12
Hypocalcaemia (Metabolism and nutrition disorders) | 99 | 141 | 27 | 30
Hypokalaemia (Metabolism and nutrition disorders) | 140 | 129 | 26 | 26
Hypomagnesaemia (Metabolism and nutrition disorders) | 52 | 39 | 7 | 9
Hypophosphataemia (Metabolism and nutrition disorders) | 48 | 59 | 15 | 12
Arthralgia (Musculoskeletal and connective tissue disorders) | 118 | 131 | 44 | 36
Back pain (Musculoskeletal and connective tissue disorders) | 181 | 194 | 46 | 56
Bone pain (Musculoskeletal and connective tissue disorders) | 105 | 99 | 16 | 13
Muscle spasms (Musculoskeletal and connective tissue disorders) | 50 | 63 | 28 | 27
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 82 | 72 | 20 | 23
Myalgia (Musculoskeletal and connective tissue disorders) | 55 | 50 | 15 | 6
Pain in extremity (Musculoskeletal and connective tissue disorders) | 138 | 127 | 29 | 28
Dizziness (Nervous system disorders) | 94 | 92 | 19 | 14
Headache (Nervous system disorders) | 88 | 100 | 12 | 19
Hypoaesthesia (Nervous system disorders) | 47 | 52 | 11 | 9
Neuropathy peripheral (Nervous system disorders) | 147 | 134 | 17 | 14
Paraesthesia (Nervous system disorders) | 73 | 70 | 12 | 11
Peripheral sensory neuropathy (Nervous system disorders) | 73 | 80 | 12 | 5
Anxiety (Psychiatric disorders) | 72 | 61 | 4 | 7
Depression (Psychiatric disorders) | 66 | 47 | 4 | 8
Insomnia (Psychiatric disorders) | 135 | 132 | 20 | 15
Cough (Respiratory, thoracic and mediastinal disorders) | 170 | 159 | 51 | 47
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 96 | 83 | 22 | 25
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 46 | 65 | 13 | 12
Alopecia (Skin and subcutaneous tissue disorders) | 48 | 56 | 0 | 4
Pruritus (Skin and subcutaneous tissue disorders) | 51 | 54 | 6 | 12
Rash (Skin and subcutaneous tissue disorders) | 102 | 132 | 17 | 17
Hypertension (Vascular disorders) | 70 | 63 | 13 | 16
Hypotension (Vascular disorders) | 39 | 50 | 6 | 7
Leukopenia (Blood and lymphatic system disorders) | 41 | 47 | 10 | 10
Abdominal pain upper (Gastrointestinal disorders) | 44 | 42 | 9 | 6
Toothache (Gastrointestinal disorders) | 45 | 50 | 27 | 16
Pain (General disorders) | 39 | 45 | 5 | 16
Influenza (Infections and infestations) | 33 | 26 | 23 | 23
Pneumonia (Infections and infestations) | 50 | 41 | 20 | 13
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 44 | 42 | 7 | 13
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 24 | 38 | 22 | 36

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.